CLINICAL TRIAL: NCT02701062
Title: AtriClip® Left Atrial Appendage Exclusion Concomitant to Structural Heart Procedures (ATLAS)
Acronym: ATLAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CP2015-2
Record Dates: First submitted 2016-02-22; First posted 2016-03-08 (Estimated); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2019-06

CONDITIONS: Post-Operative Atrial Fibrillation
Keywords: Left Atrial Appendage; Anticoagulation; CHA2DS2- VASc; HASBLED
MeSH Terms: interventions — Anticoagulation Bridge; Warfarin; Rivaroxaban; apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- LAA Exclusion with AtriClip® (Other): LAA Exclusion with AtriClip®: AtriClip® is used per label and is not experimental.
  Interventions: Device: AtriClip® Gillinov-Cosgrove™ LAA Exclusion Systems
- Medical Management (Active Comparator): Medical Management: Standard of Care Oral Anticoagulation Therapy at the discretion of the Investigator.
  Interventions: Drug: Anticoagulation Therapy

INTERVENTIONS:
Device: AtriClip® Gillinov-Cosgrove™ LAA Exclusion Systems
  Other Names: AtriClip FLEX (ACH2); AtriClip Long (LAA); AtriClip Standard (ACH1)
  Arms: LAA Exclusion with AtriClip®
Drug: Anticoagulation Therapy — Anticoagulation Therapy- Standard of Care at the discretion of the Investigator.
  Other Names: Warfarin/Coumadin; New oral anticoagulants (NOACs): dabigatran, rivaroxaban, apixaban
  Arms: Medical Management

SUMMARY:
Patients without a documented history of Atrial Fibrillation (AF) and will undergo a valve or Coronary Artery Bypass Graft (CABG) procedure with direct visual access to the Left Atrial Appendage (LAA) will be eligible to participate. Patients enrolled will be randomized 2:1 (2 with AtriClip to 1 without AtriClip. Subjects who develop Post-operative Atrial Fibrillation (POAF) and receive the AtriClip will be followed for 365 days post index procedure.

DETAILED DESCRIPTION:
Patients without a documented history of AF but who present with a CHA2DS2- VASc (congestive heart failure, hypertension, age ≥ 75 years, diabetes mellitus, stroke or transient ischemic attack (TIA), vascular disease, age 65 to 74 years, sex category) of => 2 and HASBLED (Hypertension, Abnormal Renal/Liver Function, Stroke, Bleeding History or Predisposition, Labile INR, Elderly, Drugs/Alcohol Concomitantly) of => 2 and will undergo a valve or CABG (structural heart) procedure with direct visual access to the LAA will be eligible to participate based upon the inclusion and exclusion criteria defined in this protocol. Up to 2000 patients will enroll at up to 40 sites and will be randomized 2:1 (2 with AtriClip to 1 without AtriClip. Subjects who not develop Post-operative Atrial Fibrillation (POAF) will be followed for 30 days for safety. Subjects who develop POAF and receive the AtriClip will be followed for 365 days post index procedure.

ELIGIBILITY:
Inclusion Criteria:

Patients satisfying the following criteria will be considered the screening population and will be eligible for participation:

* Age > 18 years male or female.
* Scheduled for any non-mechanical valve and/or CABG (structural heart) procedure where direct access to the LAA is expected.
* No documented preoperative AF.
* CHA2DS2-VASc score of => 2.
* HASBLED score of => 2.
* Acceptable surgical candidate, including use of general anesthesia.
* Willing and able to provide written informed consent.

Exclusion Criteria:

Patients satisfying the following criteria will not be eligible for participation:

* Redo cardiac surgery.
* Mechanical heart valve or other anticipated or current requirement for anticoagulation therapy during the post-operative (30 day) period.
* Hypercoagulability conditions that may confound the study.
* Ejection Fraction < 30.
* Left Atrium > 6 cm.
* Severe Diastolic Dysfunction.
* Requires anticoagulation therapy.
* Patient had a stroke/cerebrovascular accident (CVA) within previous 30 days prior to signing informed consent.

Intra-Operative Exclusion Criteria

* Presence of thrombus in the left atrium or LAA.
* LAA tissue is deemed friable or has significant adhesions (as evaluated by the surgeon) near or on the LAA making AtriClip placement overly risky.
* Left atrial appendage is outside the range of manufacturer's recommendations - width < 29mm or > 50mm.
* Direct visualization access is not available for AtriClip placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2016-02; Primary Completion 2019-04-26 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Gaynor, MD, Study Chair — AtriCure, Inc.
Locations (22):
- United States (22):
  - Sharp Memorial Hospital, San Diego, California
  - Stanford University, Stanford, California
  - Orlando Health Heart Institute, Orlando, Florida
  - Emory St Joseph Hospital, Atlanta, Georgia
  - St Francis Heart Hospital, Indianapolis, Indiana
  - St. Vincent Heart Center, Inc., Indianapolis, Indiana
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Maryland, Baltimore, Maryland
  - United Heart & Vascular Clinic, Saint Paul, Minnesota
  - Cardiology Associates Research, Tupelo, Mississippi
  - NYU Langone Medical Center, New York, New York
  - Mount Sinai -St. Luke's, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Christ Hospital -Linder Research Center, Cincinnati, Ohio
  - Tri-Health, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - PinnacleHealth Hospitals, Harrisburg, Pennsylvania
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Cardiovascular Surgery Clinic, Memphis, Tennessee
  - Valley Health System, Winchester, Virginia
  - Swedish Medical Center/Cherry Hill Campus, Seattle, Washington
  - Aspirus Wausau Hospital, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients without a documented history of Atrial Fibrillation (AF) but who presented with a CHA2DS2- VASc of => 2 and HASBLED of => 2 and were to undergo a valve or CABG (structural heart) procedure with direct visual access to the Left Atrial Appendage (LAA) were recruited to participate based upon the inclusion and exclusion criteria defined in the protocol. A total of 562 participants were enrolled across 23 sites. The study visits took place between February 2016 and April 2019.
Pre-assignment Details: Prior to randomization, transesophageal echocardiography (TEE) with Doppler was performed to assess for presence of thrombus. If a thrombus was present in the left atrium (LA) or LAA, the subject was not included in the study.
Groups:
- AtriClip®: LAA Exclusion with AtriClip®: AtriClip® is used per label and is not experimental.
  AtriClip® Gillinov-Cosgrove™ LAA Exclusion Systems
- No AtriClip®: Medical Management: Standard of Care Oral Anticoagulation Therapy at the discretion of the Investigator.
  Other Names:
  * Warfarin/Coumadin
  * New oral anticoagulants (NOACs): dabigatran, rivaroxaban, apixaban
  No AtriClip® used.
Period: Baseline
Arm/Group | AtriClip® | No AtriClip®
Started | 376 | 186
Completed | 376 | 186
Not Completed | 0 | 0
Period: Index Procedure
Arm/Group | AtriClip® | No AtriClip®
Started | 376 | 186
Completed | 376 | 186
Not Completed | 0 | 0
Period: Discharge
Arm/Group | AtriClip® | No AtriClip®
Started | 376 | 186
Completed | 376 | 186
Not Completed | 0 | 0
Period: 30 Day Follow-up
Arm/Group | AtriClip® | No AtriClip®
Started | 376 | 186
Completed | 366 | 183
Not Completed | 10 | 3
Period: 90 Day Follow-up
Arm/Group | AtriClip® | No AtriClip®
Started | 366 | 183
Completed | 308 | 72
Not Completed | 58 | 111
Period: 365 Day Follow-up
Arm/Group | AtriClip® | No AtriClip®
Started | 308 | 72
Completed | 294 | 69
Not Completed | 14 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AtriClip® | No AtriClip® | Total
Number analyzed (Participants) | 376 | 186 | 562
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (7.8) | 68.9 (8.7) | 69.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 50 | 163
  Male | 263 | 136 | 399
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 370 | 180 | 550
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaskan Native | 0 | 1 | 1
  Race: Asian | 5 | 2 | 7
  Race: Black or African American | 13 | 7 | 20
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Race: White | 354 | 171 | 525
  Race: Other | 3 | 3 | 6
  Race: More Than One Race | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 376 | 186 | 562
BMI (kg/m²) [Mean (Standard Deviation); unit: kg/m²] | 31.0 (5.6) | 30.0 (5.9) | 30.6 (5.7)
Risk Assessment: CHA2DS2VASc Score [Mean (Standard Deviation); unit: units on a scale] — The CHA2DS2-VASc (congestive heart failure, hypertension, age ≥ 75 years, diabetes mellitus, stroke or transient ischemic attack (TIA), vascular disease, age 65 to 74 years, sex category) score has been validated to define the risk of stroke in Atrial Fibrillation (AF) patients in numerous papers. This is a 9 point scale with 0 indicating a low risk and 9 indicating a very high risk. A CHA2DS2-VASc of >2 estimates an annual risk of stroke of between 4.5-18.2% in patients with AF.
  units on a scale | 3.4 (1.2) | 3.4 (1.1) | 3.4 (1.2)
Risk Assessment: HAS-BLED Score [Mean (Standard Deviation); unit: units on a scale] — The HAS-BLED (Hypertension, Abnormal Renal/Liver Function, Stroke, Bleeding History or Predisposition, Labile International Normalized Ratio (INR), Elderly, Drugs/Alcohol Concomitantly) score assesses the risk of major bleeding on a 9 point scale with 0 indicating a low risk and 9 indicating a very high risk.
  units on a scale | 2.8 (0.7) | 2.9 (0.6) | 2.8 (0.7)
Echocardiogram: Left Atrial Diameter (cm) [Mean (Standard Deviation); unit: cm] | 4.0 (0.7) | 3.9 (0.6) | 4.0 (0.6)
Echocardiogram: Left Atrial Diameter (cm) [Median (Full Range); unit: cm] | 3.9 [2.1 to 6.0] | 3.9 [1.9 to 5.6] | 3.9 [1.9 to 6.0]
Echocardiogram: Left Ventricular Ejection Fraction % [Mean (Standard Deviation); unit: %] | 57.3 (8.4) | 58.7 (6.9) | 57.8 (8.0)
Echocardiogram: Left Ventricular Ejection Fraction % [Median (Full Range); unit: %] | 60.0 [30.0 to 81.0] | 60.0 [35.0 to 72.0] | 60.0 [30.0 to 81.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Perioperative Complications Associated With AtriClip Placement
Description: Defined as: stroke, major bleeding that requires re-operation and/or transfusion of > 2 U packed red blood cells (PRBC), myocardial infarction (MI), or death.
Time Frame: Within any 24 hour period during the first 2 days post-index procedure
Measure: Number; unit: perioperative complications reported
Arm/Group | AtriClip®
Number analyzed (Participants) | 376
perioperative complications reported | 0

2. Secondary Outcome: Number of Subjects With Intraoperative Successful Exclusion of LAA.
Description: Successful exclusion of LAA is defined as no (0 mm) flow between LAA and LA and < 5 mm LAA remnant by intraoperative TEE with Doppler.
Time Frame: Intraoperative period
Population: Of the 376 surgical cases where placement of an AtriClip was attempted:
  * 3 AtriClip devices were not implanted
  * 2 patients could not have the intra-operative TEE imaging assessments verified post-operatively and were removed from the LAA exclusion analyses for stump and flow.
  * 1 patient that had a reported stump did not have an assessment for flow recorded.
  Therefore, 370 patients had complete data available to assess intra-operative LAA exclusion success.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AtriClip®
Number analyzed (Participants) | 370
percentage of participants
  Total Patients, No Flow and No Stump | 82.2 [77.9 to 85.9]
  Total Patients, No Flow with Stump <= 5mm | 95.4 [92.7 to 97.3]
  Total Patients, No Flow with Stump <= 10mm | 98.9 [97.3 to 99.7]

3. Secondary Outcome: Composite Event Rates Between Subjects Diagnosed With Post-operative Atrial Fibrillation (POAF) (Through 365 Days)
Description: Events to be evaluated include: Thromboembolic & Hemorrhagic Events such as cerebrovascular accident (CVA), transient ischemic attack (TIA), peripheral ischemia, hemorrhagic stroke, neurologic bleed, gastrointestinal (GI) bleeds, or other major bleeding event.
Time Frame: 365 days post index procedure
Population: Analysis includes only subjects diagnosed with POAF through 365 days.
Measure: Number; unit: percent of participants
Groups:
- AtriClip With OAC: Patients in the AtriClip group that were administered an Oral Anticoagulant (OAC) at any time following the procedure
- AtriClip Without OAC: Patients in the AtriClip group that were not administered an Oral Anticoagulant (OAC) at any time following the procedure
- Standard of Care With OAC: Patients in the No AtriClip (Standard of Care) group that were administered an Oral Anticoagulant (OAC) at any time following the procedure
- Standard of Care Without OAC: Patients in the No AtriClip (Standard of Care) group that were not administered an Oral Anticoagulant (OAC) at any time following the procedure
- Combined Standard of Care: Combined Standard of Care group with or without OAC
Arm/Group | AtriClip With OAC | AtriClip Without OAC | Standard of Care With OAC | Standard of Care Without OAC | Combined Standard of Care
Number analyzed (Participants) | 56 | 122 | 25 | 46 | 71
percent of participants | 19.6 | 8.2 | 16.0 | 6.5 | 9.9
Statistical Analysis 1: Comparison: AtriClip Without OAC vs Standard of Care With OAC; Test type: Superiority; p = 0.2593, Fisher Exact

4. Secondary Outcome: Composite Event Rates Between Subjects Not Diagnosed With POAF (Through 30 Days)
Description: as for outcome 3
Time Frame: 30 days Post-Procedure
Population: Analysis includes only subjects not diagnosed with POAF through 365 days.
Measure: Number; unit: percent of participants
Arm/Group | AtriClip With OAC | AtriClip Without OAC | Standard of Care With OAC | Standard of Care Without OAC | Combined Standard of Care
Number analyzed (Participants) | 20 | 178 | 2 | 113 | 115
percent of participants | 5.0 | 5.1 | 0.0 | 8.0 | 7.8
Statistical Analysis 1: Comparison: AtriClip Without OAC vs Standard of Care With OAC; Test type: Superiority; p = 1.000, Fisher Exact

5. Secondary Outcome: Composite Event Rates for ALL Subjects Regardless of POAF Through 365 Days
Description: as for outcome 3
Time Frame: 365 Days Post-Procedure
Measure: Number; unit: percent of participants
Groups:
- Combined AtriClip: Combined AtriClip group with or without OAC
Arm/Group | AtriClip With OAC | AtriClip Without OAC | Combined AtriClip | Standard of Care With OAC | Standard of Care Without OAC | Combined Standard of Care
Number analyzed (Participants) | 76 | 300 | 376 | 27 | 159 | 186
percent of participants | 15.8 | 6.7 | 8.5 | 14.8 | 7.5 | 8.6
Statistical Analysis 1: Comparison: AtriClip Without OAC vs Standard of Care With OAC; Test type: Superiority; p = 0.1238, Fisher Exact

6. Secondary Outcome: Healthcare Resource Utilization Variance Between Groups as Related to the Composite Events Above (Mean Values)
Description: Healthcare resource utilization variance between groups as related to hospital length-of-stay (LOS) and hospital readmissions.
Time Frame: 365 Days Post-Procedure
Population: In LOS (Total), 1 Subject removed due to incorrect date entry
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AtriClip With OAC | AtriClip Without OAC | Standard of Care With OAC | Standard of Care Without OAC
Number analyzed (Participants) | 76 | 300 | 27 | 159
days
  LOS (Total): number analyzed (Participants) | 76 | 299 | 27 | 159
  LOS (Total) | 9.1 (7.0) | 8.1 (5.2) | 8.4 (3.5) | 7.3 (4.4)
  LOS (Post-Procedure) | 7.7 (5.3) | 6.4 (3.8) | 7.7 (3.1) | 5.9 (2.7)
  Readmission LOS (per subject): number analyzed (Participants) | 9 | 11 | 2 | 4
  Readmission LOS (per subject) | 6.1 (4.1) | 4.7 (3.4) | 21.0 (18.4) | 7.0 (8.3)
Statistical Analysis 1: Comparison: AtriClip Without OAC vs Standard of Care With OAC; LOS (Total); Test type: Superiority; p = 0.6603, t-test, 2 sided
Statistical Analysis 2: Comparison: AtriClip Without OAC vs Standard of Care With OAC; LOS (Post-Procedure); Test type: Superiority; p = 0.0783, t-test, 2 sided
Statistical Analysis 3: Comparison: AtriClip Without OAC vs Standard of Care With OAC; Readmission LOS (per subject); Test type: Superiority; p = 0.4282, t-test, 2 sided

7. Secondary Outcome: Healthcare Resource Utilization Variance Between Groups as Related to the Composite Events Above (Median Values)
Description: as for outcome 6
Time Frame: 365 Days Post-Procedure
Population: In LOS (Total), 1 Subject removed due to incorrect date entry
Measure: Median (Full Range); unit: days
Arm/Group | AtriClip With OAC | AtriClip Without OAC | Standard of Care With OAC | Standard of Care Without OAC
Number analyzed (Participants) | 76 | 300 | 27 | 159
days
  LOS (Total): number analyzed (Participants) | 76 | 299 | 27 | 159
  LOS (Total) | 7.0 [3.0 to 43] | 7.0 [1.0 to 49.0] | 9.0 [3.0 to 17.0] | 6.0 [2.0 to 32.0]
  LOS (Post-Procedure) | 6.0 [3.0 to 34.0] | 5.0 [1.0 to 45.0] | 7.0 [3.0 to 12.0] | 5.0 [1.0 to 21.0]
  Readmission LOS (per subject): number analyzed (Participants) | 9 | 11 | 2 | 4
  Readmission LOS (per subject) | 5.0 [1.0 to 12.0] | 5.0 [1.0 to 12.0] | 21.0 [8.0 to 34.0] | 4.0 [1.0 to 19.0]
Statistical Analysis 1: Comparison: AtriClip Without OAC vs Standard of Care With OAC; Test type: Superiority; p = 0.6603, t-test, 2 sided
Statistical Analysis 2: Comparison: AtriClip Without OAC vs Standard of Care With OAC; LOS (Post-Procedure); Test type: Superiority; p = 0.0783, t-test, 2 sided
Statistical Analysis 3: Comparison: AtriClip Without OAC vs Standard of Care With OAC; Readmission LOS (per subject); Test type: Superiority; p = 0.4282, t-test, 2 sided

8. Secondary Outcome: Healthcare Resource Utilization Variance Between Groups as Related to the Composite Events Above (Event Rates)
Description: Specifically, reoperation for bleeding, neurologic consults for stroke or TIA, and emergency department (ED) visits.
Time Frame: 365 Days Post-Procedure
Measure: Number; unit: percentage of participants
Arm/Group | AtriClip With OAC | AtriClip Without OAC | Standard of Care With OAC | Standard of Care Without OAC
Number analyzed (Participants) | 76 | 300 | 27 | 159
percentage of participants
  Reoperation | 3.9 | 2.7 | 3.7 | 1.3
  ED Visit | 9.2 | 3.3 | 7.4 | 4.4
  Neurologic Consult | 2.6 | 2.7 | 3.7 | 4.4
  Hospital Readmission | 11.8 | 3.7 | 7.4 | 2.5
Statistical Analysis 1: Comparison: AtriClip Without OAC vs Standard of Care With OAC; Reoperation; Test type: Superiority; p = 0.5442, Fisher Exact
Statistical Analysis 2: Comparison: AtriClip Without OAC vs Standard of Care With OAC; ED Visit; Test type: Superiority; p = 0.2598, Fisher Exact
Statistical Analysis 3: Comparison: AtriClip Without OAC vs Standard of Care With OAC; Neurologic Consult; Test type: Superiority; p = 0.5442, Fisher Exact
Statistical Analysis 4: Comparison: AtriClip Without OAC vs Standard of Care With OAC; Hospital Readmission (per subject); Test type: Superiority; p = 0.2921, Fisher Exact

ADVERSE EVENTS:
Time Frame: 365 days post-procedure
Description: Subject safety was monitored throughout the course of this study by monitoring for adverse events and product complaints related to the AtriClip device. Therefore, subjects that did not receive the device were not monitored for Adverse Events. All-cause mortality was recorded for all subjects. The AtriClip device used during the index procedure for the clinical study is cleared for marketing by the FDA and was being used within the current labeling and indications for use.
Arm/Group | AtriClip® | No AtriClip®
All-Cause Mortality (participants affected / at risk) | 20/376 | 4/186
Serious Adverse Events (participants affected / at risk) | 1/376 | 0/0
Other Adverse Events (participants affected / at risk) | 1/376 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AtriClip® (N=376) | No AtriClip® (N=0)
Torsion of the heart (Cardiac disorders) | 1 (1) | 0 (0) — Unanticipated severe event that occurred post-placement, before discharge. Related to surgical technical phenomenon & the AtriClip application procedure. Medication administered & heart was untwisted during index procedure. Resolved without sequelae.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AtriClip® (N=376) | No AtriClip® (N=0)
Acute Post Pericardotomy Syndrome (Cardiac disorders) | 1 (1) | 0 (0) — Mild event that occurred post-placement, before discharge. Possibly related to the AtriClip and related to the AtriClip Device. Medication was administered. Resolved without sequelae.

LIMITATIONS AND CAVEATS:
ATLAS was an exempt post-market study therefore the use of oral anticoagulants could not be directed or standardized across the study sites. This led to a wide variation to the medical post-operative management in both the types drugs used for oral anticoagulation and dosage prescribed. Furthermore, the sample size for this feasibility study is relatively small to allow for a definitive conclusion on the impact of LAA occlusion and thromboembolic events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Before publishing or presenting, PI shall submit copies to Sponsor at least 60 days in advance. If Sponsor makes a good faith determination within such period that this release would be detrimental to its or its affiliates' intellectual property interests, PI shall refrain from publishing for another 90 days to allow Sponsor to file patent applications or take other steps to protect interests. Alternatively, these sections and/or inaccurately reported results may be redacted or modified.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT02701062/Prot_SAP_000.pdf